CLINICAL TRIAL: NCT05858086
Title: Is Postoperative Physical Therapy Clearance Necessary for Safe Home Discharge After Total Joint Arthroplasty?
Brief Title: Is Physical Therapy Clearance Before Arthroplasty Home Discharge Necessary?
Acronym: PTClearSHoT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Sumon Nandi, Clinical Professor, Chief of Adult Reconstruction, Director of Orthopaedic Research, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12
Record Dates: First submitted 2022-12-13; First posted 2023-05-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Physical Therapy; Total Joint Arthroplasty; Same-day Discharge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Postoperative Physical Therapy Clearance (Active Comparator): Patients will be evaluated and cleared by physical therapy after total joint replacement surgery prior to home discharge
  Interventions: Other: Conventional postoperative physical therapy clearance
- Preoperative Physical Therapy, Postoperative Ambulation with Nursing (Experimental): Patients will receive gait/stair training from physical therapy prior to total joint arthroplasty, then ambulate with nursing postoperatively prior to home discharge
  Interventions: Other: Novel same-day discharge protocol after total joint arthroplasty

INTERVENTIONS:
Other: Novel same-day discharge protocol after total joint arthroplasty — Preoperative gait/stair training with physical therapy, then postoperative ambulation with nursing after total joint arthroplasty
  Arms: Preoperative Physical Therapy, Postoperative Ambulation with Nursing
Other: Conventional postoperative physical therapy clearance — Physical therapy evaluation and clearance after total joint arthroplasty
  Arms: Conventional Postoperative Physical Therapy Clearance

SUMMARY:
Conventionally, physical therapy (PT) clearance is sought before total joint arthroplasty (TJA) discharge. However, PT staffing limitations may preclude same-day discharge in patients having surgery late in the day. Failed same-day discharge in eligible TJA patients results in unnecessary hospital bed occupancy, which increases costs, limits operating room throughput for patients requiring inpatient admission, and introduces risks associated with longer length-of-stay.

In collaboration with an institutional PT department, the investigators developed a protocol for discharging same-day TJA patients without postoperative PT clearance. Immediately preoperatively, PT administers gait training. Patients are then discharged home after ambulating with post-anesthesia care unit (PACU) nurses trained by PT on postoperative mobilization. This allows for the maximum number of patients discharged home, including the last patient of the day, PT staffing limitations notwithstanding. Single-institution pilot data demonstrates no increased risk of falls, emergency room (ER) visits, or readmissions with this process.

The investigators propose a prospective, controlled, multicenter study to expand on pilot data. The study aim is to assess safety of day-of-surgery preoperative PT and postoperative ambulation with PACU nursing before TJA discharge. The primary endpoint is postoperative falls, while secondary endpoints include 90-day ER visits, 90-day hospital readmissions, patient-reported outcome measures, and patient satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older
* undergo primary THA or TKA
* are eligible for same-day home discharge (friends or family available to stay at home with the patient for one week postoperatively and medically stable for discharge from PACU per anesthesia).

Exclusion Criteria:

* 90 years of age or older
* have sleep apnea (not eligible for same-day discharge)
* require overnight stay for any reason
* undergo revision THA or TKA.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of postoperative falls per patient | 6 weeks postoperatively

SECONDARY OUTCOMES:
Number of emergency room visits per patient | 90 days postoperatively
Number of hospital readmissions per patient | 90 days postoperatively
Patient satisfaction scores | 6 weeks postoperatively
  Surgical Satisfaction Questionnaire-8 (SSQ-8; range 0-100) and numeric satisfaction scale (NSS; range 0-100). Higher scores denote better outcome.
Patient reported outcome measure | 6 weeks postoperatively
  Knee Injury and Osteoarthritis Outcome Score (KOOS, JR; range 0-100). Higher scores denote better outcome.
Patient reported outcome measure | 6 weeks postoperatively
  Hip Disability and Osteoarthritis Outcome Score (HOOS, JR; range 0-100). Higher scores denote better outcome.
Patient reported outcome measure | 6 weeks postoperatively
  Patient-Reported Outcomes Measurement Information System (PROMIS; mean score 50 with standard deviation of 10). Higher scores denote more of measured domain.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - Hospital for Special Surgery, New York, New York